CLINICAL TRIAL: NCT01916356
Title: Improving Knowledge About Infertility Etiologies, Risk Factors, Treatments and Fertility Myths; an Online Educational Tool
Brief Title: Improving Knowledge About Infertility; an Online Educational Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Robert Reid, Professor, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: OBGY-241-1 6009929
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Infertility
Keywords: Infertility; Education; Risk Factors; Fertility knowledge; Fertility myths
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- educational video (Experimental): Change in participant's infertility knowledge before and after watching the educational video covering the topics of basic reproductive biology, infertility etiologies, risk factors, treatments and common myths.
  Interventions: Other: educational video

INTERVENTIONS:
Other: educational video — Educational video covering topics of basic reproductive biology, infertility etiologies, risk factors, treatments and common myths.

SUMMARY:
The purpose of this study is to determine the effectiveness of an online informational video in improving knowledge about infertility in couples experiencing problems conceiving. A pilot study will be conducted with first and second year medical students.

DETAILED DESCRIPTION:
This study is being conducted to assess how a short, online educational video changes knowledge about fertility and infertility in couples attending an infertility clinic for the first time. Participants will complete a questionnaire testing knowledge about infertility and general demographic information (age, gender, previous information sources on infertility, etc.) will be collected. Participants will then be directed to a short video on infertility. One week later, participants will return to the site to complete the infertility test questions a second time in order to test memory retention. The focus of both the questionnaire and educational video will be basic reproductive biology, infertility risk factors, etiologies and treatments and fertility myths.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 60 years
* Men between the ages of 18 and 60 years
* Booking an appointment at the infertility clinic for the first time
* Access to a computer with internet connection
* For pilot study: students must be in first or second year medical school before teaching on infertility

Exclusion Criteria:

* Previous appointment at the infertility clinic/ previous medical specialist counsel about infertility
* Completion of the study surveys after their appointment at the infertility clinic

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Mean change in total score on knowledge test | 7 days after viewing educational video
  Participants will complete an online knowledge test pre- and post-educational video. The mean change in knowledge score for each participant will be used as the primary outcome.

SECONDARY OUTCOMES:
Effect of demographic characteristics on mean change in total score on knowledge test. | 7 days after viewing educational video
  The effect of demographic variables (age, gender, education level, previous sources of information on infertility and rating of their current infertility knowledge) on infertility knowledge test scores.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Reid, M.D., Principal Investigator — Queen's University
Locations (1):
- Department of Obstetrics and Gynecology, Queen's University, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Thomson AA, Brown M, Zhang S, Stern E, Hahn PM, Reid RL. Evaluating Acquisition of Knowledge about Infertility Using a Whiteboard Video. J Obstet Gynaecol Can. 2016 Jul;38(7):646-50. doi: 10.1016/j.jogc.2016.03.010. Epub 2016 May 6. PMID 27591348